CLINICAL TRIAL: NCT03919721
Title: Phase II Field Test of Motivity.Net - Therapy Management System for Model-Based Behavioral Interventions
Brief Title: Field Test of Motivity.Net Software for Data Collection During Behavioral Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Experiad LLC (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Washington (Other); northwest behavioral associates (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Motivity-II; R44MH098476 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Autistic Disorder
Keywords: applied behavioral analysis; data collection software
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Intervention Model Description: All children enrolled in the study will already receiving ABA therapy Each tutor-child pair will have worked together regularly for at least 3 months prior to the study. Each child will have 15-20 active therapy programs, each of which will be randomly assigned to one of two sets: the experimental (Motivity-enabled) or control (therapy-as-usual). For the control set, BTs will use their existing methods, either paper-based or a competitor's data collection system. Tutors will use Motivity for 8 weeks in therapy under supervision in a single case-study pilot.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Learners receiving Applied Behavior Analysis therapy (Experimental): All children enrolled in the study will already receiving therapy. Each BT-child pair will have worked together regularly for at least 3 months prior to the study.
  Interventions: Behavioral: Applied Behavioral Analysis

INTERVENTIONS:
Behavioral: Applied Behavioral Analysis — Children are receiving Applied Behavioral Analysis therapy to treat their autism. Therapy is comprised of 15-20 discrete programs that are intended to shape specific behaviors. Tutors collect data on child's performance towards goals. For each child, some of the programs will be tracked with paper data collection methods, others will use electronic data collection. This study is to test the usefulness of the electronic data collection system to replace paper in existing interventions.

SUMMARY:
This is a study funded by a Phase II SBIR to build and test the feasibility of a new software prototype for delivering evidence-based behavioral therapy treatment for autism. The software, called Motivity.net, will be used by behavioral therapy provider groups across the country to manage the intensive data collection and analysis workflow associated with Applied Behavioral Analysis (ABA) and related therapies, which are becoming standard-of-care treatment for children with autism.

DETAILED DESCRIPTION:
This is a study funded by a Phase II SBIR to build and test the feasibility of a new software prototype for delivering evidence-based behavioral therapy treatment for autism. The software, called Motivity.net, will be used by behavioral therapy provider groups across the country to manage the intensive data collection and analysis workflow associated with Applied Behavioral Analysis (ABA) and related therapies, which are becoming standard-of-care treatment for children with autism. Experiad will conduct an 8-week within-subject pilot study of 6 BCBAs, 12 BTs and 12 children to answer product research questions about Motivity's ability to perform its intended functions, measuring the degree to which it allows interventionists to encode their models, achieve more efficient program management, improve communication, and increase responsiveness to a child's progress. Experiad will also use descriptive statistics to provide preliminary insight into the potential impact of the system on a child's performance in their ABA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Child receiving applied behavior analysis at participating institution to treat autism disorder

Exclusion Criteria:

* None

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Impact of software on number of updates to programs made by behavior analysts (intervention agility) | Data will be collected continuously from start to end of study; totals will be analyzed at the end of study (8 weeks from start date)
  Comparing the frequency of program updates between electronic programs and paper programs
Event tracking usability assessed by user ratings | Likert scale to be administered at the end of study (8 weeks from start date)
  Number of tutors who rate it highly on likert scale
Program editing efficiency as assessed by usage analysis | Time will be tracked continuously from start to end of study; totals will be analyzed at the end of study (8 weeks from start date)
  Comparison of total time spent editing electronic programs vs paper programs.
Impact of software on trial success rate | Data will be collected continuously from start to end of study; totals will be analyzed at the end of study (8 weeks from start date)
  Comparison of overall trial success rate (percent of trails meeting success threshold) in electronic administered programs compared to paper administered programs
Impact of software on trials to criterion (number of trials needed to achieve mastery) | Data will be collected continuously from start to end of study; totals will be analyzed at the end of study (8 weeks from start date)
  Comparison of trials to criterion (number of trials needed to achieve mastery) in electronic administered programs compared to paper administered programs
Impact of software on total number of targets mastered | Data will be collected continuously from start to end of study; totals will be analyzed at the end of study (8 weeks from start date)
  Comparison of total number of targets mastered in electronic administered programs compared to paper administered programs

CONTACTS AND LOCATIONS:
Overall Officials: Rex Rex, PhD, Principal Investigator — Experiad Solutions
Locations (1):
- Northwest Behavioral Associates, Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Motivity online software for use by behavioral therapists — http://www.motivity.net